CLINICAL TRIAL: NCT03070340
Title: Comparison of Breast Magnetic Resonance Imaging (MRI) and Contrast Enhanced Mammography (CEDM) to Evaluate Residual Disease Extent After Neoadjuvant Therapy (NAT)
Brief Title: Comparison of MRI and CEDM to Evaluate Treatment Response Before Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-045
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: mastectomy; breast MRI; contrast enhanced mammography; CEDM; 17-045
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast MRI and Contrast Enhanced Mammography (CEDM) (Experimental): Breast MRI and CEDM will be performed within 30 days of one another after neoadjuvant therapy
  Interventions: Diagnostic Test: Breast Magnetic Resonance Imaging (MRI); Diagnostic Test: Contrast Enhanced Mammography (CEDM)

INTERVENTIONS:
Diagnostic Test: Breast Magnetic Resonance Imaging (MRI) — All women who are scheduled for a post-NAT breast MRI and mammogram will be asked to enroll in the study. The addition of contrast to the FFDM (CEDM) would be the only intervention.
Diagnostic Test: Contrast Enhanced Mammography (CEDM) — All women who are scheduled for a post-NAT breast MRI and mammogram will be asked to enroll in the study. The addition of contrast to the FFDM (CEDM) would be the only intervention.

SUMMARY:
The purpose of this study is to compare the diagnostic accuracy of breast magnetic resonance imaging (MRI) and contrast enhanced digital mammography (CEDM) in assessing the residual disease extent in patients who have completed neoadjuvant therapy (NAT).

ELIGIBILITY:
Inclusion Criteria:

* Any woman who has completed or is nearing completion of neoadjuvant therapy for breast cancer and is scheduled for a post-NAT breast MRI and mammogram
* Surgery (mastectomy or BCT) planned within 60 days of the MRI

Exclusion Criteria:

* Women who have a contraindication to the intravenous use of iodinated contrast agent (i.e., allergy to iodinated contrast or severely impaired renal function with a creatinine level > 1.3 or eGFR ≥45)
* Known allergic reaction to gadolinium; patient may be eligible if the referring physician determines that the MRI is medically necessary and if the patient is willing to undergo pre-medication for contrast allergy
* Pregnant women
* Male patients
* Presence of non MR compatible metallic objects or metallic objects that, in the opinion of the radiologist, would make MRI a contraindication
* Known or suspected renal impairment. Requirements for GFR prior to MRI as determined by local site standard practice
* Women who have already had their standard of care post-NAT mammogram and/or breast MRI

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Compare diagnostic accuracy of breast MRI and CEDM | 1 year
  To compare the diagnostic accuracy of enhancement on MRI and CEDM in evaluating residual disease extent in women who have completed NAT prior to surgical excision

CONTACTS AND LOCATIONS:
Overall Officials: Janice Sung, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org